CLINICAL TRIAL: NCT04299802
Title: A Prospective Randomized Comparison Study on the Effects of Percutaneous Ultrasonic Tenotomy Versus Leukocyte-Rich Platelet Rich Plasma for Refractory Gluteal Tendinopathy
Brief Title: Percutaneous Ultrasonic Tenotomy Versus Platelet Rich Plasma for Gluteal Tendinopathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study not being pursued
Sponsor: Andrews Research & Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 112233
Record Dates: First submitted 2020-03-04; First posted 2020-03-09 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Gluteal Tendinitis; Trochanteric Bursitis; Tendinopathy
Keywords: Gluteal Tendinopathy; Trochanteric Bursitis; Platelet-Rich Plasma; Percutaneous Ultrasonic Tenotomy; Orthobiologics; Lateral Hip Pain
MeSH Terms: conditions — Tendinopathy | interventions — Guanfacine

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial tracking Platelet-Rich Plasma injection vs. Percutaneous Ultrasonic Tenotomy for up to 1 year
Masking Description: Unable to blind procedures as they require different types of devices, procedures and settings.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leukocyte-Rich Platelet-Rich Plasma (LR-PRP) (Active Comparator): LR-PRP will be administered via usual protocol with venous blood draw and concentration via centrifugation. The LR-PRP will be injected under ultrasound guidance into the gluteus minimus and gluteus medius tendons, enthesis and surrounding bursae.
  Interventions: Drug: Leukocyte-Rich Platelet-Rich Plasma
- Percutaneous Ultrasonic Tenotomy (Active Comparator): Percutaneous Ultrasonic Tenotomy will be administered via usual protocol within an outpatient surgical setting or in-office procedure. Patient will be anesthetized with local anesthetic and a <5mm incision will be made along the lateral hip with an #11 scalpel. A 14-G angiocath will be introduced through the defective area of the tendon down to the enthesis. Multiple passes will be made and then the percutaneous ultrasonic tenotomy device will be introduced to the defective area. No more than 5 minutes of energy cutting time will be used to address the defective area down to the enthesis, which will debride abnormal tissue but leave normal healthy tissue intact.
  Interventions: Procedure: Percutaneous Ultrasonic Tenotomy

INTERVENTIONS:
Drug: Leukocyte-Rich Platelet-Rich Plasma — LR-PRP will be a concentration of PRP with the addition of leukocytes. Studies have shown that LR-PRP is more effective in treating tendinopathy than leukocyte-poor platelet-rich plasma.
  Other Names: LR-PRP; PRP
  Arms: Leukocyte-Rich Platelet-Rich Plasma (LR-PRP)
Procedure: Percutaneous Ultrasonic Tenotomy — Discussed in Percutaneous Ultrasonic Tenotomy Arm section
  Other Names: TENEX
  Arms: Percutaneous Ultrasonic Tenotomy

SUMMARY:
The primary objective of this study is to evaluate safety and effectiveness of both a single percutaneous ultrasonic tenotomy or a single injection of LR-PRP in gluteal tendinopathy. Effectiveness will be demonstrated in a superiority trial design by comparing improvement in pain and function after a single percutaneous ultrasonic tenotomy versus a single injection of LR-PRP in refractory gluteal tendinopathy that has failed conservative management. The investigators hypothesize that both procedures will show improvement to pain and function from baseline to 24 weeks and improvement will remain at 48 weeks follow-up. The investigators propose to test this hypothesis with a series of randomized cases of gluteal tendinopathy treated with one of the proposed treatment arms and evaluate at specified intervals with validated clinical outcome measures.

DETAILED DESCRIPTION:
Aim of the Study:

To investigate the safety and effectiveness of a single percutaneous ultrasonic tenotomy procedure versus a single injection of autologous leukocyte-rich platelet rich plasma (LR-PRP) in subjects with symptomatic gluteal tendinopathy which has been refractory to conservative treatment

Hypothesis of the Study:

The hypothesis of this study is that subjects with symptomatic gluteal tendinopathy (defined as <50% partial-thickness tear of either the gluteus medius or gluteus minimus tendons on MRI or US) who receive either a single percutaneous ultrasonic tenotomy or a single injection of LR-PRP will demonstrate less pain and improved hip function compared to pre-treatment baseline.

Primary Objective:

The primary objective of this study is to evaluate safety and effectiveness of both a single percutaneous ultrasonic tenotomy or a single injection of LR-PRP in gluteal tendinopathy. Effectiveness will be demonstrated in a superiority trial design by comparing improvement in pain and function after a single percutaneous ultrasonic tenotomy versus a single injection of LR-PRP in refractory gluteal tendinopathy that has failed conservative management.

Randomization:

Subjects will be randomly assigned to the single percutaneous ultrasonic tenotomy procedure or single injection of LR-PRP arms in a 1:1 ratio.

Enrollment:

The providers from the Andrews Institute will enroll subjects into the study. 60 subjects assigned to two randomization arms will be enrolled: a single percutaneous ultrasonic tenotomy procedure arm and a single LR-PRP injection arm.

Study Duration:

Estimated Subject Enrollment Period: 36 weeks Treatment and Follow-up Period per Subject: 48 weeks

Follow-up Schedule:

Follow-up visits will occur at 2 weeks, 6 weeks, 12 weeks, 24 weeks and 48 weeks post-procedure. Visits will include physical examinations, patient-reported outcome questionnaires, medication usage, adverse event monitoring and MRIs. Follow-up phone calls will occur at 24 and 48 weeks post-procedure. Phone calls will include patient-reported outcome questionnaires, medication usage, and adverse event monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18 - 70 years of age (inclusive)
* Clinical symptoms for a minimum of three months
* Subjects have a baseline pain score of > 3
* Partial-thickness gluteal tendon tear (gluteus medius or gluteus minimus) defined as <50% partial-thickness tear of either tendon or imaging abnormalities consistent with tendinosis on a 3 Tesla MRI or diagnostic ultrasound within the last 3 months, as determined by the Investigator

Exclusion Criteria:

* Age < 18 or > 70
* Corticosteroid injection in the index gluteal bursae within the last 3 months
* Subjects who have received more than one (1) previous corticosteroid injections or percutaneous tenotomy procedure or any biologic treatment in the index gluteal bursae at any point in the past.
* Severe arthrosis of the femoral-acetabular joint
* A high-grade gluteal tendon tear (>50% partial-thickness tear)
* Previous hip surgery on the affected side
* Previous or current history of labral pathology on the affected side
* Lumbar radiculopathy impacting the index hip
* History of systemic malignant neoplasms within the last 5 years
* Malignant or local neoplasm within the last 6 months or any history of local neoplasm at the site of administration (on the affected side)
* Receiving immunosuppressive therapy
* Active regimen of chemotherapy or radiation-based treatment
* Allergy to sodium citrate or any "caine" type of local anesthetic
* Pregnancy
* Subject is currently participating in another clinical trial that has not yet completed its primary endpoint. (Non-interventional observational studies are not exclusionary.)
* Active workman's compensation case in progress

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-05-26 (Actual); Study Completion 2020-05-26 (Actual)

PRIMARY OUTCOMES:
Change in Numeric Pain Rating Scale | Baseline, 12 weeks post treatment, 48 weeks post treatment, 1 year post treatment
  Pain rating scale with a minimum score of 0 (No pain) and a maximum score of 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Change in Victorian Institute for Sport Assessment for Gluteal Tendinopathy Score | Baseline, 12 weeks post treatment, 48 weeks post treatment, 1 year post treatment
  Scores range from 0-100. Higher scores indicate less pain and better function.
Change in Hip Disability and Osteoarthritis Outcome Score | Baseline, 12 weeks post treatment, 48 weeks post treatment, 1 year post treatment
  Scores range from 0-100. 0 indicating the worst possible hip symptoms and 100 indicating no hip symptoms.
Change in Gluteal Muscle Strength | Baseline, 12 weeks post treatment, 48 weeks post treatment
  Manual muscle strength will be assessed by an investigator. The scale used will range from 0-5. Lower scores indicate less strength.

OTHER OUTCOMES:
Change in Visual Analog Scale for Procedure Satisfaction | Baseline, 24 weeks post treatment, 48 weeks post treatment
  A VAS for satisfaction is a horizontal line of 100-mm long. At the beginning and at the end, there are two descriptors representing extremes of satisfaction (i.e. no satisfaction and extreme satisfaction). The patient will make a vertical mark on the 100-mm line. The measurement in millimetres will be converted to the same number of points ranging from 0 to 100 points.

CONTACTS AND LOCATIONS:
Overall Officials: James Andrews, MD, Study Chair — Andrews Research & Education Foundation

IPD SHARING:
Plan to Share IPD: No
No HPI will be disclosed to anyone not involved with the study. The data will be published at the completion of the study and will be publicly available for consumption.

REFERENCES:
- [Result] Jacobson JA, Yablon CM, Henning PT, Kazmers IS, Urquhart A, Hallstrom B, Bedi A, Parameswaran A. Greater Trochanteric Pain Syndrome: Percutaneous Tendon Fenestration Versus Platelet-Rich Plasma Injection for Treatment of Gluteal Tendinosis. J Ultrasound Med. 2016 Nov;35(11):2413-2420. doi: 10.7863/ultra.15.11046. Epub 2016 Sep 23. PMID 27663654
- [Result] Borg-Stein J, Osoria HL, Hayano T. Regenerative Sports Medicine: Past, Present, and Future (Adapted From the PASSOR Legacy Award Presentation; AAPMR; October 2016). PM R. 2018 Oct;10(10):1083-1105. doi: 10.1016/j.pmrj.2018.07.003. Epub 2018 Jul 19. PMID 30031963
- [Result] Wu PI, Diaz R, Borg-Stein J. Platelet-Rich Plasma. Phys Med Rehabil Clin N Am. 2016 Nov;27(4):825-853. doi: 10.1016/j.pmr.2016.06.002. PMID 27788903
- [Result] Fitzpatrick J, Bulsara MK, O'Donnell J, McCrory PR, Zheng MH. The Effectiveness of Platelet-Rich Plasma Injections in Gluteal Tendinopathy: A Randomized, Double-Blind Controlled Trial Comparing a Single Platelet-Rich Plasma Injection With a Single Corticosteroid Injection. Am J Sports Med. 2018 Mar;46(4):933-939. doi: 10.1177/0363546517745525. Epub 2018 Jan 2. PMID 29293361
- [Result] Fitzpatrick J, Bulsara M, Zheng MH. The Effectiveness of Platelet-Rich Plasma in the Treatment of Tendinopathy: A Meta-analysis of Randomized Controlled Clinical Trials. Am J Sports Med. 2017 Jan;45(1):226-233. doi: 10.1177/0363546516643716. Epub 2016 Jul 21. PMID 27268111
- [Result] Lee JJ, Harrison JR, Boachie-Adjei K, Vargas E, Moley PJ. Platelet-Rich Plasma Injections With Needle Tenotomy for Gluteus Medius Tendinopathy: A Registry Study With Prospective Follow-up. Orthop J Sports Med. 2016 Nov 9;4(11):2325967116671692. doi: 10.1177/2325967116671692. eCollection 2016 Nov. PMID 27868077
- [Result] Neph A, Onishi K, Wang JH. Myths and Facts of In-Office Regenerative Procedures for Tendinopathy. Am J Phys Med Rehabil. 2019 Jun;98(6):500-511. doi: 10.1097/PHM.0000000000001097. PMID 30433886
- [Result] Morrey, Bernard F.
- [Result] Barnes DE, Beckley JM, Smith J. Percutaneous ultrasonic tenotomy for chronic elbow tendinosis: a prospective study. J Shoulder Elbow Surg. 2015 Jan;24(1):67-73. doi: 10.1016/j.jse.2014.07.017. Epub 2014 Oct 8. PMID 25306494